CLINICAL TRIAL: NCT00877422
Title: Vitamin D Supplementation Prevents Pneumonia in Institutionalized Elderly Subjects
Brief Title: Vitamin D Supplementation Prevents Elderly Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tohoku University (Other)
Responsible Party: Takashi Ohrui/MD,PhD, Institute of Development, Aging and Cancer, Tohoku University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IDAC-VD-01; KAKENHI 20390285
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Bacterial Pneumonia
Keywords: vitamin deficiency
MeSH Terms: conditions — Pneumonia, Bacterial; Avitaminosis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (No Intervention): Group A is identified as serum vitamin D level more than 16 ng/dl.
- Group B (Active Comparator): Group B is identified as serum vitamin D level less than 16 ng/dl and is supplemented with vitamin D3.
  Interventions: Dietary Supplement: Vitamin D3
- Group C (No Intervention): Group C is identified as serum vitamin D less than 16 ng/dl and is not supplemented with vitamin D3.

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Group A and Group C are followed without drugs and Group B is followed with vitamin D3.
  Arms: Group B

SUMMARY:
Pneumonia is the fourth leading cause of death and frequently occurs in institutionalized elderly people in Japan. Recently, several clinical and experimental studies have reported the importance of vitamin D in the regulation of immune functions and its deficiency is associated with susceptibility to some infections. In the present study, the investigators hypothesize that deficiency of serum vitamin D is associated with development of pneumonia, and supplementation of vitamin D may lower the incidence of pneumonia and prolong survival in institutionalized elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are more than 65 years old and were resident in the facility for at least 6 months.
* Subjects have no conditions known to interfere with vitamin D metabolism.

Exclusion Criteria:

* Subjects are excluded if they have:

  * renal failure
  * hepatic failure
  * hyper- or hypo-parathyroidism
  * HIV infection, or malignant diseases
* Subjects are also excluded if they are taking corticosteroid, thiazide diuretics, or supplementary vitamins.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-08

PRIMARY OUTCOMES:
prevalence of pneumonia | one year

SECONDARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Arai, MD, Study Chair — Department of Geriatrics and Gerontology, Tohoku University
Locations (1):
- Institute of Development, Aging and Cancer, Tohoku University, 1-1,Seiryo-machi,Aoba-ku,Sendai, Japan